CLINICAL TRIAL: NCT04557579
Title: Comparison of Quality of Vision After Bifocal and Extended Depth of Focus Intraocular Lens Implantation
Status: Completed | Type: Observational
Sponsor: Taipei Nobel Eye Clinic (Other)
Responsible Party: Principal Investigator, Chao-Kai Chang, Dean, Nobel Eye Institute, Taipei Nobel Eye Clinic
Other Study IDs: 001
Record Dates: First submitted 2020-08-27; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Intraocular Lens

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bifocal group: Patients in bifocal group implanted with Restor +2.5D IOL (Alcon, Fort Worth, TX, USA) in bilateral eyes
  Interventions: Procedure: Clear corneal phacoemulsification and IOL implantation
- Extended depth of focus group: Patients in extended depth of focus group implanted with EDOF Symfony IOL (AMO, Santa Ana, CA, USA) in bilateral eyes
  Interventions: Procedure: Clear corneal phacoemulsification and IOL implantation
- Monofocal group: Patients in monofocal group implanted with Sensar AR40e IOL (AMO, Santa Ana, CA, USA) in bilateral eyes
  Interventions: Procedure: Clear corneal phacoemulsification and IOL implantation

INTERVENTIONS:
Procedure: Clear corneal phacoemulsification and IOL implantation — Clear corneal phacoemulsification and IOL implantation were performed by 2 surgeons (Chao-Kai Chang and Hung-Yuan Lin) by using an identical technique to minimize differences in surgically induced aberrations between groups. The surgical process involved topical anesthesia, a 3-step clear corneal incision (2.75 mm) at 180° (temporal in both eyes), a 5.0-mm continuous curvilinear capsulorhexis, phacoemulsification using the stop-and-chop technique, IOL implantation with an injector, IOL centration, and a sutureless incision. The study IOL models include EDOF Symfony IOL (AMO, Santa Ana, CA, USA), bifocal Restor +2.5D IOL (Alcon, Fort Worth, TX, USA), and monofocal Sensar AR40e IOL (AMO, Santa Ana, CA, USA).

SUMMARY:
To compare the visual performance of the extended depth of focus (EDOF) intraocular lens (IOL) to bifocal and spherical monofocal IOL

DETAILED DESCRIPTION:
This study was conducted from 2018 to 2020. This study included patients who were with presence of cataract in both eyes, age between 50 and 80 years, and corrected distance visual acuity (CDVA) of both eyes under 20/40. Phacoemulsification cataract surgery was arranged for both eyes for all patients. The study groups of IOL models include EDOF Symfony IOL (AMO, Santa Ana, CA, USA), bifocal Restor +2.5D IOL (Alcon, Fort Worth, TX, USA), and monofocal Sensar AR40e IOL (AMO, Santa Ana, CA, USA). The patients were routinely examined preoperatively as well as 1 month after surgery for far and near visual acuity (in LogMAR unit). Contrast sensitivity, wavefront aberration and quality of vision questionnaire was measured at the 1-month postoperative visit. These aforementioned outcomes were recorded and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* presence of cataract in both eyes
* age between 50 and 80 years
* CDVA of both eyes under 20/40
* Phacoemulsification cataract surgery was arranged for both eyes

Exclusion Criteria:

* complicated cataract
* corneal opacities or irregularities
* corneal astigmatism > 1.5 diopter
* dry eye (Schirmer's test I ≤ 5mm)
* amblyopia
* anisometropia
* surgical complications such as posterior capsular bag rupture or vitreous loss
* IOL tilt or decentration
* coexisting ocular pathologies
* glaucoma
* non-dilating pupil
* history of intraocular surgery, laser therapy, or retinopathy
* optic nerve or macular diseases
* refusal or unable to maintain follow-up.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted from 2018 to 2020 in the Taipei Nobel Eye Clinic and Universal Eye Center ophthalmology clinic. The research protocol was explained to all prospective participants, after which they provided written informed consent before participating. The study was approved by the Ethics Committee of Chunghua Christian Hospital, and the protocol accorded with the tenets of the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Ophthalmic examinations | 1 month after surgery.
  far uncorrected visual acuity(UCVA) and corrected distance visual acuity (CDVA), near UCVA in LogMAR unit
Wavefront examination | at the 1-month postoperative visit
  Wavefront analysis was performed only at the 1-month postoperative visit with an AMO WaveScan Hartmann-Shack sensor (Santa Clara, CA, USA). The wavefront maps were analyzed using a 6-mm pupil diameter and a Zernike polynomial expansion up to the sixth-order of Zernike coefficients. Higher order aberrations including RMS errors of horizontal coma aberration (Z 3,1), spherical aberration (4,0), trefoil aberration and the higher order aberrations were assessed.
Contrast sensitivity | at the 1-month postoperative visit
  CS was also measured at the 1-month postoperative visit using the Vector Vision CSV-1000 (Greenville, OH, USA) chart. All subjects were tested at the recommended distance of 8 feet. The CSV-1000 consists of a series of circular achromatic sine-wave patches having a 1.5-in. diameter and comprising 4 rows, each corresponding to one of 4 spatial frequencies: 3, 6, 12, and 18 cycles per degree (cpd). We selected 3, 6 and 12 cpd for analysis.
Questionnaire | at the 1-month postoperative visit
  Subjective QoV was evaluated using a questionnaire adopted from a near-activity 19-item questionnaire and the NEI-RQL-42. Our questionnaire contains 11 questions and the subscales include far vision, diurnal fluctuation, glare and halos, spectacle dependence, near vision, and intermediate vision. In general, questionnaires were completed without assistance; however, on the patient's request, explanations of the questions were provided.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Kai Chang, Ph.D., Principal Investigator — Taipei Nobel Eye Clinic
Locations (1):
- Taipei Nobel Eye Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calladine D, Evans JR, Shah S, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD003169. doi: 10.1002/14651858.CD003169.pub3. PMID 22972061
- [Background] Kohnen T, Nuijts R, Levy P, Haefliger E, Alfonso JF. Visual function after bilateral implantation of apodized diffractive aspheric multifocal intraocular lenses with a +3.0 D addition. J Cataract Refract Surg. 2009 Dec;35(12):2062-9. doi: 10.1016/j.jcrs.2009.08.013. PMID 19969209
- [Background] Thibos LN, Ye M, Zhang X, Bradley A. The chromatic eye: a new reduced-eye model of ocular chromatic aberration in humans. Appl Opt. 1992 Jul 1;31(19):3594-600. doi: 10.1364/AO.31.003594. PMID 20725330
- [Background] Perez-Merino P, Dorronsoro C, Llorente L, Duran S, Jimenez-Alfaro I, Marcos S. In vivo chromatic aberration in eyes implanted with intraocular lenses. Invest Ophthalmol Vis Sci. 2013 Apr 12;54(4):2654-61. doi: 10.1167/iovs.13-11912. PMID 23493299
- [Background] Weeber HA, Piers PA. Theoretical performance of intraocular lenses correcting both spherical and chromatic aberration. J Refract Surg. 2012 Jan;28(1):48-52. doi: 10.3928/1081597X-20111103-01. Epub 2011 Nov 10. PMID 22074466
- [Background] Denoyer A, Le Lez ML, Majzoub S, Pisella PJ. Quality of vision after cataract surgery after Tecnis Z9000 intraocular lens implantation: effect of contrast sensitivity and wavefront aberration improvements on the quality of daily vision. J Cataract Refract Surg. 2007 Feb;33(2):210-6. doi: 10.1016/j.jcrs.2006.10.035. PMID 17276260